CLINICAL TRIAL: NCT06667843
Title: Smart Nutrition, Healthier Communities: A Digital Therapeutic Strategy for Early Obesity Intervention
Brief Title: Smart Nutrition, Healthier Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Stjørdal Municipally (Unknown); Lifeness AS (Unknown); National patient organization (LFO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 774938
Record Dates: First submitted 2024-10-15; First posted 2024-10-31 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Methods

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard follow-up at respective Healthy Lives Center with the addition of a digital therapeutic app with a full lifestyle program, including daily logging, tasks, articles and general information and possibility for digital communication with their healthcare provider.
  Interventions: Behavioral: Lifestyle Management; Device: Intervention
- Control (Experimental): Standard follow-up at respective Healthy Lives Center, including daily logging in the digital therapeutic app.
  Interventions: Behavioral: Lifestyle Management; Device: Control

INTERVENTIONS:
Behavioral: Lifestyle Management — Behavioral intervention for lifestyle change
Device: Intervention — Full access to DTx function in the app, and digital follow up/communication with helthcare professionals at the Healthy Lives Center
  Arms: Intervention
Device: Control — Basic access to the app (daily logging functions). No digital follow up or communication with healthcare professionals at the Healthy Lives Center.
  Arms: Control

SUMMARY:
The project investigates the effect of the health app Lifeness as a digital therapeutic (DTx) and follow-up tool in a municipal setting at a regional Healthy Lives Center in central Norway (Frisklivssentralen Værnesregionen), targeting early intervention for overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤27kg/m2 or obesity measured by waist circumference, current weight stability, motivated to lifestyle change using mobile apps, access to smartphone with 5G. Living in the municipallies covered by the Værnes region of central Norway.

Exclusion Criteria:

* previous bariatric surgery, use of anti-obesity drugs, pregnancy, current or present cancer diagnosis,substance abuse or psychiatric diagnosis (such as eating disorders), or other conditions that can hinder physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Body weight, and weight circumference, will be measured with standard proceduress (medically approved digital Seca scale (kg), and standard measuring band (cm)) wearing light clothing at baseline and after 12 weeks.

SECONDARY OUTCOMES:
Eating behavior and hedonic appetite | 12 weeks
  Validated quistionaires assessing hedonic appetite and eating behavior will be measured at baseline and after 12 weeks: Dutch Eating Behavior Questionnaire (DEBQ), Three Factor Eating Questonnaire (TFEQ), and the Power of Food Scale (PFS).
Weight related quality of life | 12 weeks
  A validated quistionaire assessing weight-related quality of life (IWQOL-Lite) will be handed out at baseline and after 12 weeks

OTHER OUTCOMES:
Feasability | 12 weeks
  Engagement in the app will be evaluated by monitoring the participants check-in streaks and progress in the DTx programme during the intervention. Usability and feasbility for both study participants and healthcare professionals will be evaluted through a standardized validation form at the end of the 12 week intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Frisklivssentralen Værnesregionen, Stjørdal, Trøndelag
  - Norwegian University of Science and Technology, Trondheim, Trøndelag

IPD SHARING:
Plan to Share IPD: Yes
Collected data at baseline and w12 (anthropometrics, BMI, eating behavior and quality of life) can be shared upon request

REFERENCES:
- [Derived] Aukan MI, Larsen MA, Melan TI, Salvesen OO. Beyond weight loss: digital therapeutic for behavioral change and psychological well-being for individuals with overweight and obesity in a primary healthcare setting-A randomized controlled pilot study. Front Digit Health. 2025 Sep 16;7:1671649. doi: 10.3389/fdgth.2025.1671649. eCollection 2025. PMID 41035564